CLINICAL TRIAL: NCT06338228
Title: A New Decisional Tree for the Management of Acetabular Fractures : Monocentric Observational Study
Acronym: FANAD
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A02458-37
Record Dates: First submitted 2024-02-14; First posted 2024-03-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Management of Acetabular Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients managed for Acetabular fracture: collect the data for all the patients managed and operated on between 01/01/2020 AND 31/01/2022 for Acetabular fracture

SUMMARY:
Acetabular fractures are challenging fractures to treat. Many fracture patterns occur, in a deep anatomical area surrounded by numerous vascular and nervous elements, generally in a polytraumatic context . A reduction with less than 2 mm of incongruence is generally considered acceptable, limiting post-operative osteoarthritis that could rapidly require total hip arthroplasty. Due to the long learning curve, this surgery is limited to large reference centers

. In the last twenty years, the main series published in the literature are small series due to the rarity of the fractures and their trauma context (loss of follow-up, polytrauma patients…). The large variety of fracture patterns according to the Letournel classification creates a spread in patient distribution and decreases the power of statistical analysis. That is the reason why big series are rare and only a few of them allow significant conclusions . The other studies are meta-analyses with their limitations

The lack of consensus makes it difficult to interpret the results between series, so the investigators developed a decision tree to address this knowledge gap.

The aim of this study is to assess and compare the results of a decisional tree for acetabular fracture in a large cohort of patients from a well-known experimental trauma center.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient at the time of injury
* Acetabular fracture
* Pre-operative standard X-ray image
* Pre-operative CT image
* Post-operative X-ray standard image (AP-alar and obturator views)
* Post-operative CT scan.
* Willingness and ability to participate in the study

Exclusion Criteria:

* Ipsilateral fracture femoral and/or associated pelvic ring fracture (Floating Hip C or B)
* Pregnant, lactating women
* Subject under administrative or judicial supervision

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients managed between 01/01/2020 and 01/01/2023 for an acetabular fracture in our trauma center are included in this single-center retrospective study.
  The epidemiological data, the pre-operative management, the fracture patterns according to the Letournel and AO/OTA classification, the operative data and the radiological criteria (X-rays and CT scans) are retrospectively collected and analyzed.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
The main objective of the study is to evaluate and compare the results of a decision tree for the management of acetabulum fractures (also called acetabulum) in a large cohort of patients from the trauma center at Grenoble University Hospital | 1 year
  Clinical results according to the Postel-Merle d'Aubigné score (PMA)

SECONDARY OUTCOMES:
Define the prognostic factors associated with poor clinical outcomes and total hip replacement surgery | 1 year
  Prognostic factors from operative data
Compare clinical and radiological findings with the literature | 1 year
  Clinical outcomes according to Harris Hip Score(HHS)
Compare clinical and radiological findings with the literature | 1 year
  Clinical outcomes according to Oxford-12 HIP score (OXFORD HIP)
Compare clinical and radiological findings with the literature | 1 year
  Clinical outcomes according to MAJEED SCORES
Compare clinical and radiological findings with the literature | 1 year
  Clinical outcomes according to NUMERIC PAIN SCALE ( from 0-to10) 0 no pain 10 worst possible pain
Compare clinical and radiological findings with the literature | 1 year
  Clinical outcomes according to radiological scores
Propose a new assessment of the traumatic hip joint based on PROMs (Patient Reported Outcomes Measures) via a dedicated digital application (Orthense by Digikare) | 1 year
  Epidemiological data based on PROMs (Patient Reported Outcomes Measures) via a dedicated digital application (Orthense by Digikare)
Evaluation of Outcomes and Complications of Early Weight Bearing in Older Adults | 1 year
  Complications intra-operative and postoperative (including complications of early weight bearing)

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi PI BOUDISSA, Pr, Principal Investigator — Grenoble Alpes University Hospital
Locations (1):
- Grenoble Alpes University Hospital,La tronche, Grenoble, France

REFERENCES:
- [Background] JUDET R, JUDET J, LETOURNEL E. FRACTURES OF THE ACETABULUM: CLASSIFICATION AND SURGICAL APPROACHES FOR OPEN REDUCTION. PRELIMINARY REPORT. J Bone Joint Surg Am. 1964 Dec;46:1615-46. No abstract available. PMID 14239854
- [Background] Matta JM, Anderson LM, Epstein HC, Hendricks P. Fractures of the acetabulum. A retrospective analysis. Clin Orthop Relat Res. 1986 Apr;(205):230-40. PMID 3698382
- [Background] Matta JM, Merritt PO. Displaced acetabular fractures. Clin Orthop Relat Res. 1988 May;(230):83-97. PMID 3365902
- [Background] Letournel E. Acetabulum fractures: classification and management. Clin Orthop Relat Res. 1980 Sep;(151):81-106. PMID 7418327
- [Background] Negrin LL, Seligson D. Results of 167 consecutive cases of acetabular fractures using the Kocher-Langenbeck approach: a case series. J Orthop Surg Res. 2017 Apr 26;12(1):66. doi: 10.1186/s13018-017-0563-6. PMID 28446184
- [Background] Kreder HJ, Rozen N, Borkhoff CM, Laflamme YG, McKee MD, Schemitsch EH, Stephen DJ. Determinants of functional outcome after simple and complex acetabular fractures involving the posterior wall. J Bone Joint Surg Br. 2006 Jun;88(6):776-82. doi: 10.1302/0301-620X.88B6.17342. PMID 16720773
- [Background] Wang XJ, Lu Li, Zhang ZH, Su YX, Guo XS, Wei XC, Wei L. Ilioinguinal approach versus Stoppa approach for open reduction and internal fixation in the treatment of displaced acetabular fractures: A systematic review and meta-analysis. Chin J Traumatol. 2017 Aug;20(4):229-234. doi: 10.1016/j.cjtee.2017.01.005. Epub 2017 Jun 19. PMID 28709737
- [Background] Shazar N, Eshed I, Ackshota N, Hershkovich O, Khazanov A, Herman A. Comparison of acetabular fracture reduction quality by the ilioinguinal or the anterior intrapelvic (modified Rives-Stoppa) surgical approaches. J Orthop Trauma. 2014 Jun;28(6):313-9. doi: 10.1097/01.bot.0000435627.56658.53. PMID 24100918
- [Background] Giannoudis PV, Grotz MR, Papakostidis C, Dinopoulos H. Operative treatment of displaced fractures of the acetabulum. A meta-analysis. J Bone Joint Surg Br. 2005 Jan;87(1):2-9. PMID 15686228
- [Background] Mears DC, Velyvis JH, Chang CP. Displaced acetabular fractures managed operatively: indicators of outcome. Clin Orthop Relat Res. 2003 Feb;(407):173-86. doi: 10.1097/00003086-200302000-00026. PMID 12567145
- [Background] Murphy D, Kaliszer M, Rice J, McElwain JP. Outcome after acetabular fracture. Prognostic factors and their inter-relationships. Injury. 2003 Jul;34(7):512-7. doi: 10.1016/s0020-1383(02)00349-2. PMID 12832177
- [Background] Tannast M, Najibi S, Matta JM. Two to twenty-year survivorship of the hip in 810 patients with operatively treated acetabular fractures. J Bone Joint Surg Am. 2012 Sep 5;94(17):1559-67. doi: 10.2106/JBJS.K.00444. PMID 22992846
- [Background] Boudissa M, Ruatti S, Kerschbaumer G, Milaire M, Merloz P, Tonetti J. Part 2: outcome of acetabular fractures and associated prognostic factors-a ten-year retrospective study of one hundred and fifty six operated cases with open reduction and internal fixation. Int Orthop. 2016 Oct;40(10):2151-2156. doi: 10.1007/s00264-015-3070-6. Epub 2015 Dec 21. PMID 26686672
- [Background] Boudissa M, Francony F, Kerschbaumer G, Ruatti S, Milaire M, Merloz P, Tonetti J. Epidemiology and treatment of acetabular fractures in a level-1 trauma centre: Retrospective study of 414 patients over 10 years. Orthop Traumatol Surg Res. 2017 May;103(3):335-339. doi: 10.1016/j.otsr.2017.01.004. Epub 2017 Feb 22. PMID 28235575